CLINICAL TRIAL: NCT00406887
Title: Phase 3 Confirmatory Study of 0.05% Difluprednate Ophthalmic Emulsion in the Treatment of Anterior Uveitis (Including Panuveitis).
Brief Title: Study of Difluprednate Ophthalmic Emulsion in the Treatment of Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJE2079/3-01-PC
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Anterior Uveitis; Panuveitis
MeSH Terms: conditions — Uveitis, Anterior; Panuveitis

INTERVENTIONS:
Drug: Difluprednate Ophthalmic Emulsion

SUMMARY:
The purpose of this phase 3 confirmatory study is to determine if difluprednate ophthalmic emulsion is effective in the treatment of treatment of uveitis.

DETAILED DESCRIPTION:
The objective of this phase 3 study is to assess the efficacy and safety of 0.05% difluprednate ophthalmic emulsion (DFBA) in patients with endogenous anterior uveitis, in comparison with 0.1% betamethasone sodium phosphate ophthalmic solution (BP).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with endogenous anterior uveitis or panuveitis
* Patients with 10 - 49 anterior chamber cells within one field of the anterior chamber as observed by slit lamp microscopy (criterion for rating of signs 2 or 3)
* Patients aged ‰1425 years (on the day of obtaining informed consent) who were able to accurately express their own symptoms
* Patients provided written informed consent prior to initiation of the study

Exclusion Criteria:

* Patients who did not meet all of the above inclusion criteria
* Patients received systemic administration of any corticosteroid or immunosuppressive drug within the past 1 week prior to instillation of the investigational product
* Patients received topical injection of any corticosteroid in eyes prior to instillation of the investigational product (Solution formulation: within the past 1 week, depot: within the past 2 weeks)
* Patients received systemic administration of any non-steroidal anti-inflammatory drug or antiphlogistic enzyme within the past 3 days prior to instillation of the investigational product
* Patients received instillation of any corticosteroid, non-steroidal anti-inflammatory drug or antiphlogistic enzyme within 12 hours prior to instillation of the investigational product
* Patients with glaucoma or ocular hypertension
* Patients with corneal abrasion or ulcer
* Patients with any confirmed or suspected viral, bacterial or fungal keratoconjunctival disease
* Patients with allergy to similar drugs such as other corticosteroids
* Patients requiring use of contact lens during the study period
* Women who are or might be pregnant, or lactating women
* Patients participating in another clinical study within the past 3 months before initiation of the present study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140
Dates: Start 2002-08; Study Completion 2003-11

PRIMARY OUTCOMES:
The difference from the baseline in anterior chamber cell score on Day 14
was compared between the two groups.

SECONDARY OUTCOMES:
The differences from the baseline in anterior chamber cell score on Days 3 and 7
were compared between the two groups.
The numbers of patients with an anterior chamber cell score of 0 on Days 7 and
14 were compared between the two groups.
The differences from the baseline in total sign and symptom scores on Days 3, 7
and 14 were compared between the two groups.
The numbers of patients with an anterior chamber cell score of 1 or less on Days
3, 7 and 14 were compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeaki Ohno, PhD, Principal Investigator — Department of Ophthalmology and Visual Science, Graduate School of Medicine, Hokkaido University